CLINICAL TRIAL: NCT04924127
Title: Exploring the Feasibility of the Molecular Pathology Model of Patients With Glioma Via Retrospective Research
Brief Title: Molecular Pathology Research Project of Glioma
Status: Completed | Type: Observational
Sponsor: Jinsong Wu (Other)
Responsible Party: Sponsor-Investigator, Jinsong Wu, Prof., Huashan Hospital
Organization: Huashan Hospital (Other)
Other Study IDs: KY2019-539
Record Dates: First submitted 2021-05-23; First posted 2021-06-11 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Glioma, Malignant
Keywords: Molecular pathology
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Discovery cohort: Retrospective frozen tissue and paired peripheral blood samples were obtained from the Huashan Glioma Biobank between October 2010 and August 2018. A total of 753 patients diagnosed with supratentorial diffuse glioma (WHO grade 2-4) aged 18-80 years were selected for the study.
  Interventions: Diagnostic Test: Detection of IDH and TERT mutation
- Validation cohort: From January to July 2021, 223 frozen tissue samples were retrieved from the Huashan Glioma Biobank. In addition, 107 frozen tumor samples were used to assess the detection accuracy of the IDH and TERTp mutation rapid test. The accuracy of this qPCR-based rapid test was further confirmed by Sanger and targeted sequencing.
  Interventions: Diagnostic Test: Detection of IDH and TERT mutation

INTERVENTIONS:
Diagnostic Test: Detection of IDH and TERT mutation — Detection of IDH and TERT mutation using frozen glioma tissues

SUMMARY:
Evaluate the diagnostic value of TERT promoter mutation in differ glioma subtypes and expend the application of the diagnostic algorithm to surgical practice

DETAILED DESCRIPTION:
A total of 976 gliomas were enrolled in this study. First, in order to evaluate the diagnostic value of TERT promoter mutation in differ glioma subtypes, we conducted a retrospective cohort study included 753 frozen tissue samples of patients with different grades of glioma. According to WHO CNS5, all recommended alteration including IDH, 1p/19q, TERT, EGFRamp and 7+/10- were profiled using multiple approaches and a permanent diagnosis was obtained for each patient. Exploring the feasibility of the molecular pathology model of patients with glioma via retrospective research. Compare with the existing molecular pathology system, analyze the combination of IDH and TERT mutations and the feasibility of stratifying the prognosis of patients with glioma.

Moreover, to expend the application of the diagnostic algorithm to surgical practice, we developed a fast detection assay that could detect hotspot somatic mutations in IDH and TERT within 25 minutes and can discriminate TERT and IDH mutations from wild-type alleles with a minimum variant allele frequency (VAF) of 0.2% and 0.5%, respectively. We further validate the simplified diagnostic algorithm on frozen tissue of 223 patients with glioma in another retrospective cohort and performed this assay to evaluate the accuracy of the rapid assay.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Glioma
* Glioma patient with long-term follow-up data and intact clinical data

Exclusion Criteria:

* Glioma patient without Informed Consent Form
* Glioma patient without long-term follow-up data or intact clinical data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glioma patient from Huashan Hospital with Informed Consent Form
Sampling Method: Non-Probability Sample
Enrollment: 976 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Evaluate the diagnostic value of TERT promoter mutation in differ glioma subtypes | through study completion, an average of 1 week
  According to WHO CNS5, all recommended alteration including IDH, 1p/19q, TERT, EGFRamp and 7+/10- were profiled using multiple approaches and a permanent diagnosis was obtained for each patient. Exploring the feasibility of the molecular pathology model of patients with glioma
Derivation and validation of a simplified diagnostic scheme | through study completion, an average of 1 week
  Derivation of a simplified diagnostic scheme based on IDH and TERT promoter (TERTp) mutations combined with histology and evaluation of its feasibility of stratifying the prognosis of patients with glioma when comparing with WHO CNS5 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-song Wu, MD & PhD, Study Chair — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, Jingan District, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu J, Wu S, Cao D, Xiong Z, Zhang J, Zou Y, Wu Z, Nie Y, Luo C, Yao Y, Song Y, Jiao Y, Chen H, Ma H, Kang D, Mao Y, Yan H. Rapid diagnosis of adult-type diffuse glioma using a layered scheme. BMC Med. 2025 Jun 2;23(1):325. doi: 10.1186/s12916-025-04124-9. PMID 40457320